CLINICAL TRIAL: NCT00801164
Title: Exploratory Study of Iocide Oral Rinse in a Diabetic Population
Acronym: Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biomedical Development Corporation (Industry)
Collaborators: Methodist Healthcare Ministries of South Texas (Unknown); Foundation Of Collaborative Unique Science (FOCUS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSC20080508H
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Type 2; Periodontitis
Keywords: Diabetes Type 2; Periodontitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Frio Oral Rinse (Experimental): Prescription Mouth Rinse. Rinse with 15ml twice daily then expectorate.
  Interventions: Drug: Frio Mouth Rinse
- Placebo (Experimental): Prescription Mouth Rinse. Rinse with 15ml twice daily then expectorate.
  Interventions: Drug: Frio Mouth Rinse Placebo

INTERVENTIONS:
Drug: Frio Mouth Rinse Placebo — Prescription Mouth Rinse. Rinse with 15ml twice daily then expectorate.
  Arms: Placebo
Drug: Frio Mouth Rinse — Prescription Mouth Rinse. Rinse with 15ml twice daily then expectorate.
  Arms: Frio Oral Rinse

SUMMARY:
The goals of this exploratory study are to 1)examine an investigational oral rinse as an adjunctive agent to scaling and root planing in treating chronic periodontitis in a periodontitis-susceptible diabetes population, and 2) evaluate its effect on glycemic control and biomarkers of systemic inflammation.

DETAILED DESCRIPTION:
This double-blind prospective pilot study will evaluate the effects of an investigational oral rinse as an adjunctive agent to non-surgical periodontal intervention for patients with type 2 diabetes mellitus. Approximately thirty (30) adult (35 years or older) patients with type 2 diabetes mellitus with untreated chronic periodontitis of moderate or worse severity will be enrolled in the 6-month study to provide 24 evaluable subjects (12 per group). All subjects enrolled in the trial will receive standard periodontal therapy including scaling and root planing (SRP). Half will be randomized to receive the investigational oral rinse adjunctively twice daily; the other half will receive placebo rinse twice daily. Study participants will be treated with either Iocide or placebo rinse for the first 90 days of the study only. Follow up examinations will be performed at six months. Evaluation of biological markers associated with systemic inflammation and diabetes will be performed at baseline, three months, and six months. The primary study outcome is clinical measurement of chronic periodontitis (gingival index, bleeding on probing, probing depth, clinical attachment level). Secondary outcomes are change in HbA1c and markers of systemic inflammation measured by serum C-reactive protein, plasma TNF-a, and IL-6.

ELIGIBILITY:
Inclusion Criteria:

1. Have self-reported type 2 diabetes of more than three months duration.
2. A current HbA1c value between 7.0% and 12%.
3. Report no change in diabetes-related medications during the three months prior to enrollment.
4. Be at least 35 years of age.
5. Have at least 16 natural teeth.
6. Have moderate to severe chronic periodontitis, defined by loss of clinical attachment of >5 mm on two seperate teeth, and no treatment within six months.
7. Able and willing to comply with study requirements including following instructions on study treatment and returning for follow-up visits as required by the protocol
8. Have full understanding of all elements of, and signature and dating of the written informed consent prior to the initiation of protocol specified procedures
9. Females with childbearing potential must have a negative pregnancy test before and during the study period. Sexually active females must be using an effective form of birth control. These methods include oral contraceptives ("the pill"), an intrauterine device (IUD), levonogestrol implants (Norplant®), medroxyprogesterone acetate injections (Depo-provera®) or contraceptive foam with a condom.

Exclusion Criteria:

1. History, or current evidence, of any significant acute or chronic medical or psychiatric condition that, in the opinion of the Investigator, would render examination difficult or invalid or prevent the subject from active study participation
2. TPOab positive
3. Baseline serum level of TSH <0.35 or >5.5
4. Treatment with antibiotic within the three (3) month period prior to the screening examination
5. Presence of valvular disease, prosthetic implant, or any other systemic condition requiring antibiotic premedication
6. History of thyroid disease
7. Purported sensitivity or allergy to iodine
8. Known sensitivity or allergy to shellfish
9. History of autoimmune disease, or chronic infections such as HIV or hepatitis
10. History of cardiovascular disease (heart attack or procedure within the past three months, stroke or history/treatment for transient ischemic attacks in the past three months, or documented history of pulmonary embolus in past six months), unstable angina pectoris or angina pectoris at rest,
11. History of renal disease: serum creatinine exceeding 1.4 mg/dl (women) or 1.5 mg/dl (men), or currently receiving dialysis.
12. Gross oral pathology (periodontal disease, rampant caries, tissue damage created by poor oral care or treatment, soft or hard tissue tumors) that, in the opinion of the Investigator, could alter the treatment needs during the study
13. Current signs or symptoms of mucosal tissue ulcerations or inflammation, or canker sores
14. Presence of orthodontic appliances or any removable appliance that impinges on the oral tissues being assessed
15. History of or current alcohol abuse that, in the opinion of the Investigator, could influence the outcome of the study
16. History of, or current drug abuse
17. Use of concomitant medication that, in the opinion of the Investigator, might interfere with the outcome of the study (e.g. antibiotics, immuno-suppressants, steroids, or therapeutic doses of non-steroidal anti-inflammatory agents, phenytoin, calcium antagonists, cyclosporine or coumadin)
18. Concomitant therapy with another investigational drug or device without prior approval from the Sponsor within four weeks prior to Visit 2 (Study Day 1)
19. Concomitant endodontic or periodontal therapy other than prophylaxis in the past six (6) months
20. Females with childbearing potential with a positive pregnancy test, pregnant or nursing mothers, suspected pregnancy, or intention to become pregnant during the study
21. Residence in the same household as a subject already enrolled in the study (inclusion may create blinding and/or compliance issues)
22. Unable and unwilling to comply with the informed consent process, to meet study requirements including following instructions on study treatment, and to return for follow-up visits as required by the protocol.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary study endpoints are periodontal evaluation including clinical attachment level, pocket depth, plaque index, suppuration and gingival index score. | 6 Months

SECONDARY OUTCOMES:
Secondary endpoints include glycated hemoglobin A1c (HbA1c) and systemic biomarkers (LPS, TNF-a, CRP, IL-6, serum insulin and glucose). Tertiary outcome measures include staining, calculus, opportunistic Candida infection, and patient satisfaction. | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W. Oates, DMD, Ph.D., Principal Investigator — University of Texas
Locations (1):
- The University of Texas Health Science Center at San Antonio, Dental School, San Antonio, Texas, United States